CLINICAL TRIAL: NCT05335603
Title: Fatty Liver Library (FALL): a Prospective Cohort Study Evaluating the Characteristics of Chronic Liver Diseases Associated With Hepatic Steatosis
Brief Title: An Observational Study Evaluating Patients With Chronic Liver Diseases Associated With Hepatic Steatosis
Acronym: FALL
Status: Recruiting | Type: Observational
Sponsor: University of Copenhagen (Other)
Collaborators: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Nicolai Jacob Wewer Albrechtsen, Associate professor, University of Copenhagen
Other Study IDs: FALL
Record Dates: First submitted 2022-04-12; First posted 2022-04-19 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Chronic Liver Disease
Keywords: non-alcoholic fatty liver disease; non-alcoholic steatohepatitis; steatosis; autoimmune hepatitis; primary biliary cholangitis; primary sclerosing cholangitis; haemochromatosis; alfa-1-antitrypsin deficiency; chronic pancreatitis; chronic liver disease; inflammatory bowel disease; OMICS; Mass spectrometry
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver; Hepatitis, Autoimmune; Liver Cirrhosis, Biliary; Cholangitis, Sclerosing; Hemochromatosis; Pancreatitis, Chronic; Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Liver tissue, plasma, serum, whole blood.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hepatic steatosis may cause inflammation and fibrosis within the liver potentially leading to end-stage liver disease cirrhosis, liver failure and death. The condition is associated with several other chronic liver diseases like autoimmune hepatitis, primary biliary cholangitis, primary sclerosing cholangitis, hereditary hemochromatosis and alpha-1-antitrypsin deficiency and may also develop secondary to other diseases like inflammatory bowel disease and chronic pancreatitis. Diagnosing chronic liver diseases can be challenging and treatment may be limited. In-depth phenotyping at a tissue level may generate insight into the underlying pathophysiology of diseases and furthermore identify common as well as specific diagnostic biomarkers and future treatment targets of the diseases. We therefore undertake a study that evaluates patients with chronic liver diseases associated with hepatic steatosis.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients/healthy control participants (age 18 or above) who can give their informed consent
* Suspected liver disease:
* non-alcoholic steatohepatitis
* alcoholic steatohepatitis
* autoimmune hepatitis
* primary biliary cholangitis
* primary sclerosing cholangitis
* inflammatory bowel disease
* polycystic ovary syndrome
* hereditary haemochromatosis
* chronic pancreatitis
* cystic fibrosis
* alpha-1 antitrypsin deficiency

Exclusion Criteria:

Patients with:

* malignant diseases
* viral hepatitis
* human immunodeficiency virus
* contraindications to liver biopsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Potentially eligible patients will be identified and recruited among those referred with suspected liver disease at the outpatient clinic at the Gastro Unit, Copenhagen University Hospital Hvidovre, Denmark. Healthy control participants will be recruited through advertisements at forsoegsperson.dk and posters. Posters will be mounted in neutral places at Copenhagen University Hospital Hvidovre and at neutral places at the Panum Institute. Copenhagen University Hospital Hvidovre is a large regional hospital with more than 3500 employees and the Panum Institute is a large building complex in Copenhagen, Denmark that houses the Faculty of Health and Medical Sciences.
Sampling Method: Non-Probability Sample
Enrollment: 335 (Estimated)
Dates: Start 2020-08-24 (Actual); Primary Completion 2036-08 (Estimated); Study Completion 2036-08 (Estimated)

PRIMARY OUTCOMES:
Identification and validation of a diagnostic classifier enabling discrimination of chronic liver diseases. | 10 years
  OMICS based analyses on plasma and liver tissue

SECONDARY OUTCOMES:
To identify any metabolic disturbances within chronic liver diseases | Plasma obtained at time point 0 min, 15 min, 30 min, 45 min, 60 min, 90 min, 120 min.
  Collection of plasma during an oral glucose tolerance test measuring pancreatic and gut hormones

OTHER OUTCOMES:
Fibrosis stage of the liver | 10 years
  Non-invasive scoring systems (e.g. Fibroscan, Fib-4)

CONTACTS AND LOCATIONS:
Overall Officials: Lise L Gluud, Professor, Principal Investigator — Hvidovre University Hospital; Nicolai J Wewer Albrechtsen, MD, PhD, Principal Investigator — NNF Center for Protein Research
Locations (1):
- Hvidovre University Hospital, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jensen AH, Ytting H, Nielsen AB, Werge MP, Rashu EB, Hetland LE, Thing M, Nabilou P, Burisch J, Junker AE, Hobolth L, Mortensen C, Tofteng F, Bendtsen F, Moller S, Vyberg M, Serizawa RR, Winther-Sorensen M, Kellemann JS, Gluud LL, Wewer Albrechtsen NJ. Diagnostics of Autoimmune Hepatitis Enabled by Non-Invasive Clinical Proteomics. Aliment Pharmacol Ther. 2025 Nov;62(9):901-919. doi: 10.1111/apt.70273. Epub 2025 Jul 17. PMID 40671462